CLINICAL TRIAL: NCT01618188
Title: A Trial Investigating the Pharmacodynamic Properties of NN1218 in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-3978; U1111-1126-0900 (Other: WHO); 2011-005796-16 (EudraCT Number)
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Formulation A (Experimental)
  Interventions: Drug: Faster-acting insulin aspart
- Formulation B (Experimental)
  Interventions: Drug: Faster-acting insulin aspart
- Insulin Aspart (Active Comparator)
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: Faster-acting insulin aspart — A single dose of 0.2 U/kg body weight for subcutaneous (s.c., under the skin) administration.
  Other Names: NN1218
  Arms: Formulation A; Formulation B
Drug: insulin aspart — A single dose of 0.2 U/kg body weight for subcutaneous (s.c., under the skin) administration.
  Arms: Insulin Aspart

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the pharmacodynamic properties (the effect of the investigated drug on the body) of NN1218 in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus for more than 12 months
* Treated with multiple daily insulin injections or continuous subcutaneous insulin infusion for more than 12 months
* Body mass index (BMI) between 18.0-28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to trial start
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine substitute products during the inpatient period

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2012-06-11 (Actual); Primary Completion 2012-09-07 (Actual); Study Completion 2012-09-07 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve | From 0 to 2 hours

SECONDARY OUTCOMES:
Area under the glucose infusion rate curve | From 0 to 12 hours
Maximum glucose infusion rate | Within 0 to 12 hours after dosing
Time to maximum glucose infusion rate | Within 0 to 12 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Background] Heise T, Hovelmann U, Brondsted L, Adrian CL, Nosek L, Haahr H. Faster-acting insulin aspart: earlier onset of appearance and greater early pharmacokinetic and pharmacodynamic effects than insulin aspart. Diabetes Obes Metab. 2015 Jul;17(7):682-8. doi: 10.1111/dom.12468. Epub 2015 May 8. PMID 25846340
- [Background] Haahr H, Hövelmann U, Brøndsted L, Adrian CL, Nosek L, Heise T. Higher Early Insulin Exposure and Greater Early Glucose-lowering Effect with Faster-acting Insulin Aspart in Patients with Type 1 Diabetes Mellitus (T1DM). Diabetes 2014; 63 ((Suppl 1)): A233 (abstract 910-P)
- [Background] Heise T, Pieber TR, Danne T, Erichsen L, Haahr H. Faster Onset and Greater Early Exposure and Glucose-Lowering Effect with Faster-Acting Insulin Aspart vs. Insulin Aspart: A Pooled Analysis in Subjects with Type 1 Diabetes. Diabetes. 2016; Suppl. 1: A239. doi:10.2337/db16-861-1374 http://dx.doi.org/10.2337/db16-861-1374
- [Result] Haahr H, Pieber TR, Mathieu C, Gondolf T, Shiramoto M, Erichsen L, Heise T. Clinical Pharmacology of Fast-Acting Insulin Aspart Versus Insulin Aspart Measured as Free or Total Insulin Aspart and the Relation to Anti-Insulin Aspart Antibody Levels in Subjects with Type 1 Diabetes Mellitus. Clin Pharmacokinet. 2019 May;58(5):639-649. doi: 10.1007/s40262-018-0718-6. PMID 30402720
- [Derived] Heise T, Pieber TR, Danne T, Erichsen L, Haahr H. A Pooled Analysis of Clinical Pharmacology Trials Investigating the Pharmacokinetic and Pharmacodynamic Characteristics of Fast-Acting Insulin Aspart in Adults with Type 1 Diabetes. Clin Pharmacokinet. 2017 May;56(5):551-559. doi: 10.1007/s40262-017-0514-8. PMID 28205039
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com